CLINICAL TRIAL: NCT00567372
Title: POSTERIOR SUB-TENON'S CAPSULE INJECTION OF BEVACIZUMAB FOR TREATMENT OF DIFFUSE DIABETIC MACULAR EDEMA
Brief Title: POSTERIOR SUB-TENON'S Avastin
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00922
Record Dates: First submitted 2007-11-30; First posted 2007-12-04 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Diffuse Diabetic Macular Edema
Keywords: Diffuse diabetic macular edema; sub-tenon; Bevacizumab
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bevacizumab (Sub-tenon´s injection) — a single posterior sub-tenon's capsule injection of bevacizumab (2.5 mg /0.1ml)

SUMMARY:
Posterior sub-tenon's injection of bevacizumab decreased diffuse diabetic macular edema

ELIGIBILITY:
Inclusion Criteria:

Patients with diffuse diabetic macular edema non-proliferative diabetic retinopathy Maculat thickness ≥250 μ BCVA ≥ 20/400 Without any treatment

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2008-11 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
macular volume | baseline, 3,6 and 12 weeks

SECONDARY OUTCOMES:
macular thickness | baseline,3,6 and 12 weeks
best corrected visual acuity | baseline, 3,6 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Vera, MD, Principal Investigator — Asociación para Evitar la Ceguera en Mexico; Hugo Quiroz-Mercado, MD, Principal Investigator — Denver Health Medical Center; Adai Pérez-Montesinos, MD, Principal Investigator — Asociación para Evitar la Ceguera en Mexico
Locations (1):
- Asociación para Evitar la Ceguera en Mexico, Mexico City, Mexico City, Mexico